CLINICAL TRIAL: NCT01476189
Title: A Repeat Dose PK Study Investigating the Extent of Paracetamol Absorption From Two Sustained Release Paracetamol Formulations
Brief Title: A Study to Compare to the Pharmacokinetic Profile of Two Paracetamol Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A2750607
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Subjects
Keywords: pharmacokinetic; paracetamol; Healthy volunteer; steady state

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental paracetamol formulation (Experimental): test formulation
  Interventions: Drug: Experimental paracetamol formulation
- Marketed paracetamol (Active Comparator): Marketed paracetamol
  Interventions: Drug: Marketed paracetamol
- Higher dose marketed paracetamol (Active Comparator): higher dose marketed paracetamol
  Interventions: Drug: Higher dose marketed paracetamol

INTERVENTIONS:
Drug: Experimental paracetamol formulation — experimental
  Arms: Experimental paracetamol formulation
Drug: Marketed paracetamol — Marketed paracetamol
  Arms: Marketed paracetamol
Drug: Higher dose marketed paracetamol — Higher dose marketed paracetamol
  Arms: Higher dose marketed paracetamol

SUMMARY:
A repeat dose pharmacokinetic study investigating two paracetamol formulations

ELIGIBILITY:
Inclusion Criteria:

* Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination.

Exclusion Criteria:

* Subject does not agree to refrain from alcohol consumption for the 10-day period prior to visit 2 and throughout the study.
* Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
* Current (within 14 days of screening) or regular use of any prescription, over-the-counter drugs including paracetamol/acetaminophen, herbal medicine or drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to dosing (e.g. barbiturates, theophylline, cimetidine, or erythromycin), excluding prescription birth control, if applicable.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence as measured by Area Under the Curve (AUC) | last 24 hours of dosing

SECONDARY OUTCOMES:
Time duration at or above minimal therapeutic plasma paracetamol concentration | last 24 hours of dosing
To assess pharmacokinetic parameters (Cmax, AUC, Tmax and Kel) | last 24 hours of dosing
Adverse events | Baseline to 72 hours post dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- MDS Pharma Services NEBRASKA, Lincoln, Nebraska, United States